CLINICAL TRIAL: NCT00105599
Title: Effectiveness of the FairCare System for Patients With Advanced Illness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CHI 99-071
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Terminal Care; Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: End of life care coordination; Procedure: FairCare System

INTERVENTIONS:
Behavioral: End of life care coordination
Procedure: FairCare System

SUMMARY:
This study of the FairCare Program (FC) is designed to address end of life (EOL) care delivery issues by reducing barriers to effective EOL care among health care providers, family members, surrogates, and Chronic Heart Failure (CHF) patients using a comprehensive, multi-pronged approach delivered by a care coordinator and supported by an interdisciplinary team.

DETAILED DESCRIPTION:
Background:

This study of the FairCare Program (FC) is designed to address end of life (EOL) care delivery issues by reducing barriers to effective EOL care among health care providers, family members, surrogates, and Chronic Heart Failure (CHF) patients using a comprehensive, multi-pronged approach delivered by a care coordinator and supported by an interdisciplinary team.

Objectives:

Evaluate the impact of FC on: 1) improving the quality of life (QOL) and health care delivery for CHF patients with advanced illness, (i.e. ejection fractions of 35% or less, or assessed as level III or IV on the NYS Heart Association Classification System); 2) addressing their fears about dying; 3) increasing their use of Advance Directives (ADs); and 4) improving provider compliance with ADs. Also, describe trends that may occur in disease-specific QOL, survival, and health care use and cost.

Methods:

The study employs a randomized control group design. There are two treatment arms, the FC treatment condition, and the usual care (UC) control condition. Assessments for improving quality of life (QOL), and quality of care delivery are taken at baseline, and at three and six months. Assessments of AD use, i.e. frequency of formulation and documentation of ADs, are taken at baseline, three and six months at one year and 18 months. Because data about compliance with ADs and utilization and cost may not be fully comprehensive until patients' deaths, to maximize the sample size for these variables, and hence the power of the study to detect difference in these outcomes, data on compliance with ADs will be collected in the final year of the study, and data on utilization and cost will be aggregated in monthly intervals and collected from baseline to 18 months. One year of VA pre-intervention health care utilization and cost data will also be collected to assess baseline utilization and to control for any pre-existing differences in the propensity of patients to use health care services. Also, an intention to treat methodology will be used during data analyses.

Status:

The study ends 9-30-04, data for VA cost, Medicare cost, consistency of medical care with patient preferences, and survival, are being collected and analyzed for the final report.

ELIGIBILITY:
Inclusion Criteria:

Ejection fraction 35% or less and classification at level 3 or 4 of the New York State Heart Classification System and surrogates of patients meeting this criteria.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mollie Shulan, MD, Principal Investigator — Albany VA Medical Center Samuel S. Stratton, Albany, NY
Locations (1):
- Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York, United States